CLINICAL TRIAL: NCT01093053
Title: A Randomized Controlled Study of Mind-Body Skills Groups for Treatment of War Zone Stress in Military and Veteran Populations
Brief Title: Mind-Body Skills Groups for the Treatment of War Zone Stress in Military and Veteran Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Mind-Body Medicine (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); Southeast Louisiana Veterans Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, James S. Gordon, M.D., Founder and Director, The Center for Mind-Body Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08144040
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2014-01

CONDITIONS: Stress Disorders, Post Traumatic; Brain Injuries; Depressive Disorder; Anxiety Disorders; Anger
Keywords: Mind-Body Therapies
MeSH Terms: conditions — Combat Disorders; Brain Injuries; Depressive Disorder; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mind-Body Skills Groups (Experimental)
  Interventions: Behavioral: Mind-Body Skills Groups
- Standard Treatment (Active Comparator)
  Interventions: Other: Standard Treatment

INTERVENTIONS:
Behavioral: Mind-Body Skills Groups — The mind-body skills group program teaches participants how to do meditation, guided imagery, breathing techniques, and biofeedback. These mind-body techniques are taught and practiced in small groups of 8 to 10 people and also contain an element of social support.
  Arms: Mind-Body Skills Groups
Other: Standard Treatment — May include individual or group psychotherapy consisting of cognitive behavioral therapy or present-centered (i.e. unrelated to mindfulness) psychotherapy as well as medication management. Medications for depression, anxiety, and sleep disorders are the most commonly used in standard treatment.
  Arms: Standard Treatment

SUMMARY:
The purpose of this study is to determine whether participation in mind-body skills groups by veterans who have experienced a stressful war-related situation and have symptoms of posttraumatic stress disorder (PTSD), will improve symptoms of PTSD, depression and anxiety, reduce anger, improve quality of life, quality of sleep and result in posttraumatic growth (a positive change that people can experience when they have been in a traumatic situation).

DETAILED DESCRIPTION:
The study will be a randomized controlled study where participants will be randomly selected to either participate in the mind-body skills program and to answer questionnaires before and after the program and again 6 months later or, if they are not randomized to the mind-body skills group program, they will answer the questionnaires during the same time periods without participating in the program. Both groups will also continue their medical treatment as usual. The mind-body skills group intervention consists of groups of 8-10 participants. Two formats will be offered. (1) A 2 hour group session once a week for 10 weeks or (2) Weekend groups which will be run on alternating Saturdays, with a 2 hour session in the morning and another 2 hour session in the afternoon. The groups will be run for a total of 5 Saturday sessions. Additional "reunion" groups will be held at 1 month, 3 months, and 6 months in order to reinforce skills and to provide continuing social support.

ELIGIBILITY:
Inclusion Criteria:

* having experienced a deployment-related criterion A stressor and reporting post deployment stress symptoms which include: clinically diagnosed posttraumatic stress disorder (PTSD), or subthreshold PTSD symptoms
* comorbid conditions may also include mild traumatic brain injury, or clinically significant levels of depression or anxiety.

Exclusion Criteria:

* current uncontrolled psychotic or bipolar disorder
* significant cognitive impairment
* moderate or severe TBI
* substance dependence
* suicidal or homicidal ideation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
PTSD checklist - military version | Baseline; 12 weeks; 20 weeks
  The PTSD checklist contains 17 items corresponding to the DSM-IV criteria for PTSD. Past month symptom severity is indicated using a 5 point scale.

SECONDARY OUTCOMES:
State-Trait Anger Expression Inventory-2 | Baseline;12 weeks; 20 weeks
  This is a 57 item consisting of a 4 point scale that measures the intensity of anger as an emotional state at a particular time (State Anger) and how often angry feelings are experienced over time as a personality trait (Trait Anger). There are 4 additional subscales which measure the outward expression of anger (Anger Expression-Out), holding or suppressing angry feelings (Anger Expression-In); controlling angry feelings by preventing the outward expression of anger (Anger Control-Out); and controlling anger feeling by calming down (Anger Control-In)
The Pittsburgh Sleep Quality Index | Baseline;12 weeks; 20 weeks
  This 9 item questionnaire using a 4 point scale measures seven areas of sleep: subjective sleep quality, sleep latency, sleep duration, habitual seep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction.
The Patient Health Questionnaire-9 | Baseline;12 weeks; 20 weeks
  The Patient Health Questionnaire-9 is a 9 item self-report measure and is a widely used screening tool for depression.
State-Trait Anxiety Inventory | Baseline; 12 weeks; 20 weeks
  The State anxiety subscale will be used. It has 20 questions and uses a 4 point scale.
The Posttraumatic Growth Inventory | Baseline;12 weeks; 20 weeks
  The Posttraumatic Growth Inventory measures positive change that people can experience when they have been in a traumatic situation. It is a 21 item self report scale that includes five subscales: relating to others, new possibilities, personal strength, spiritual challenge, and appreciation of life.
The Medical Outcomes Study Short Form SF-36 | Baseline; 12 weeks; 20 weeks
  The SF-36 has 36 questions and measures functional status in eight dimensions: physical functioning, social functioning, role functioning-physical, role functioning-emotional, vitality, mental health, bodily pain, and general health perception.
The Inventory of Functional Impairment | Baseline;12 weeks; 20 weeks
  The Inventory of Functional Impairment is an 87-item self-report measure designed to assess multiple dimensions of functional impairment experienced by active duty service members and veterans.

CONTACTS AND LOCATIONS:
Overall Officials: James S Gordon, MD, Principal Investigator — The Center for Mind-Body Medicine
Locations (1):
- Southeast Louisiana Veterans Healthcare System, New Orleans, Louisiana, United States